CLINICAL TRIAL: NCT02219178
Title: A Phase II Study of the Efficacy and Safety of Lenalidomide, Subcutaneous Bortezomib, and Dexamethasone Combination Therapy for Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Study of the Efficacy and Safety of RsqVD Combination Therapy for Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 13-17; 2013-005008-32 (EudraCT Number)
Record Dates: First submitted 2014-08-11; First posted 2014-08-18 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RsqVD (Experimental): Oral lenalidomide 25mg days 1 - 14 of 21 day schedule Subcutaneous bortezomib 1.3mg/m2 days 1, 4, 8, 11 of 21 day schedule Oral dexamethasone 20mg on days 1, 2, 4, 5, 8, 9, 11, 12 of 21 day schedule
  Interventions: Drug: lenalidomide; Drug: Subcutaneous bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: lenalidomide — 25mg days 1 - 14 of 21 day schedule
  Other Names: Revlimid
Drug: Subcutaneous bortezomib — 1.3mg/m2 days 1, 4, 8, 11 of 21 day schedule
  Other Names: Velcade
Drug: Dexamethasone — 20mg on days 1, 2, 4, 5, 8, 9, 11, 12 of 21 day schedule
  Other Names: Decadron

SUMMARY:
This study aims to evaluate the overall response rate after 4 cycles and the best response to induction therapy with combination of lenalidomide, subcutaneous bortezomib, and dexamethasone (RsqVD) in patients with newly diagnosed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a diagnosis of symptomatic MM, according to International Myeloma Foundation 2003 Diagnostic Criteria:

   * Clonal plasma cells > 10% on bone marrow biopsy
   * A monoclonal protein (paraprotein) in either serum or urine ( except in the cases of non-secretory myeloma).

   If no monoclonal protein is detected (non-secretory disease), then ≥ 30% monoclonal bone marrow plasma cells and/or a biopsy-proven plasmacytoma required.
   * Evidence of end-organ damage felt related to the plasma cell disorder related organ or tissue impairment (ROTI), commonly referred to by the acronym 'CRAB':

     * Hypercalcaemia: serum calcium (corrected for albumin) > 10.5mg/sL/>2.65mmol/L or upper limit of normal
     * Renal insufficiency defined as serum creatinine > 2mg/sL/177μmol/L
     * Anaemia: Normochromic, normocytic with a haemoglobin value > 2g/dL below the lower limit of normal or a haemoglobin < 10g/dL
     * Bone lesions (lytic lesions, severe osteopenia or pathologic fractures) as shown by CT scan and/or skeletal survey
2. Patient has received no prior treatment with any systemic therapy for the treatment of multiple myeloma.

   * Prior treatment of hypercalcaemia or spinal cord compression with corticosteroids does not disqualify the patient (the dose should not exceed the equivalent of 160 mg of dexamethasone in a 2 week period)
   * Bisphosphonates are permitted
   * Patients treated with local radiotherapy with or without concomitant exposure to steroids, for pain control or management of cord/nerve root compression, are eligible. Two weeks must have lapsed since last date of radiotherapy, which is recommended to be a limited field. Patients who require concurrent radiotherapy should have entry to the protocol deferred until the radiotherapy is completed and 2 weeks have passed since the last date of therapy.
3. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
4. Age ≥ 18 years at the time of signing Informed Consent
5. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Lenalidomide Pregnancy Prevention Risk Management Plan. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mlU/mL 10 to14 days prior to therapy and repeated again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by Lenalidomide Pregnancy Prevention Risk Management Plan) and must either commit to complete abstinence from heterosexual contact or begin TWO acceptable methods of birth control, one highly effective method and one additional effective (barrier) method, AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must practice complete abstinence or agree to use a condom during sexual contact with a FCBP even if they have had a successful vasectomy. All study participants must be registered into the mandatory Lenalidomide Pregnancy Prevention Risk Management Plan, and be willing and able to comply with the requirements of the Lenalidomide Pregnancy Prevention Risk Management Plan.*A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e. has had menses at any time during the preceding 24 consecutive months)
6. All necessary baseline studies for determining eligibility must be obtained within 21 days prior to enrolment
7. Subject has an ECOG performance status of < 2 or Karnofsky performance status of ≥ 60 (Appendix E).
8. Subject must be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Patient has ≥ Grade 2 peripheral neuropathy on clinical examination within 14 days before enrolment
2. Renal insufficiency (serum creatinine levels > 2.5 mg/dL/221μmol/L, calculated creatinine clearance with Cockcroft-Gault formula (see Appendix G) < 45 ml/min)
3. Subjects with evidence of mucosal or internal bleeding and/or platelet refractory (i.e. unable to maintain a platelet count 50,000 cells/mm3)
4. Subjects with an absolute neutrophil count (ANC) < 1000 cells/mm3. Growth factors may not be used to meet ANC eligibility criteria
5. Subjects with a haemoglobin < 8.0 g/dL
6. AST (SGOT) and ALT (SGPT) > 2 x ULN, bilirubin levels 1.5 ULN
7. Concomitant therapy medications that include corticosteroids (except as indicated in inclusion criteria)
8. Myocardial infarction within 6 months prior to enrolment or has New York Heart Association (NYHA) Class III or IV heart failure (Appendix G), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
9. Clinically relevant active infection requiring treatment (antibiotics, antivirals, antifungals)
10. Any serious co-morbid condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study.
11. Female subject is pregnant or breast-feeding
12. Serious psychiatric illness or addiction likely to interfere with participation in this clinical study
13. Uncontrolled diabetes mellitus
14. Contraindication to any required concomitant drugs or supportive therapies including hypersensitivity to all anticoagulation and antiplatelet options or hypersensitivity to acyclovir or similar anti-viral drug. History of allergic reaction/hypersensitivity attributed to compounds containing boron, mannitol, polysorbate 80 or sodium citrate dehydrate
15. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes)
16. Known seropositive for or active HIV infection or active hepatitis B or C viral infection. Patients who are seropositive because of hepatitis B virus vaccine are eligible
17. Known intolerance to steroid therapy
18. Patient has hypersensitivity to bortezomib, boron, or mannitol
19. Diagnosed or treated for another malignancy within 2 years of enrolment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
20. Participation in clinical trials with other anti-myeloma investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial
21. Radiation therapy within 2 weeks before randomization. Enrolment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 2 weeks have elapsed since the last date of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2019-10-31 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall response rate (ORR) after 4 induction cycles | After 4 cycles (84 days)
  To evaluate the overall response rate (ORR) after 4 induction cycles and the best response to induction therapy with the combination of lenalidomide, subcutaneous (SQ) bortezomib, and dexamethasone (RsqVD) in patients with newly diagnosed multiple myeloma.

SECONDARY OUTCOMES:
a) To evaluate the rate and severity of Peripheral Neuropathy (PN) of SQ bortezomib in combination with lenalidomide, and dexamethasone after the 4th and after the final cycle of induction therapy. | After 4 cycles (84 days)
  Evaluate the rate and severity of Peripheral Neuropathy of SQ bortezomib in combination with lenalidomide, and dexamethasone after the 4th and after the final cycle of induction therapy
Progression of disease | Duration of the study, expected to be approximately 3 years
  Evaluate the time to progression
Progression free survival | Duration of the study, expected to be approximately 3 years
  Evaluate progression free survival
Duration of response | Duration of the study, expected to be approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Gorman, Dr, Principal Investigator — Mater Misericordiae University Hospital
Locations (8):
- Ireland (8):
  - University Hospital Waterford, Waterford, Co Waterford
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - Midlands Regional Hospital, Tullamore

REFERENCES:
- [Derived] O'Gorman P, Laubach JP, O'Dwyer ME, Krawczyk J, Yee AJ, Gilligan O, Cahill MR, Rosenblatt J, Quinn J, Murphy PT, DiPietro H, Perera MR, Crotty GM, Cummings K, Hayden PJ, Browne P, Savell A, O'Leary HM, O'Keeffe D, Masone K, Hennessy BJ, Guerrero Garcia T, Scott K, Saeed K, Bianchi G, Dowling P, Tierney C, Richardson PG. Phase 2 studies of lenalidomide, subcutaneous bortezomib, and dexamethasone as induction therapy in patients with newly diagnosed multiple myeloma. Am J Hematol. 2022 May;97(5):562-573. doi: 10.1002/ajh.26491. Epub 2022 Feb 18. PMID 35132679